CLINICAL TRIAL: NCT04172415
Title: Current Procedural Sedation Practices for Adults and Children in a Canadian Community Emergency Department
Brief Title: Current Procedural Sedation Practices in a Canadian Community Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Amber Graystone (Other)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor-Investigator, Amber Graystone, Principle Investigator, Niagara Health System
Organization: Niagara Health System (Other)
Other Study IDs: 7148-C
Record Dates: First submitted 2019-10-29; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Conscious Sedation
Keywords: Procedural Sedation; Chart Review

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective cohort: Patients that received procedural sedation in a community Emergency Department.
  Interventions: Other: Retrospective cohort

INTERVENTIONS:
Other: Retrospective cohort — Chart Review

SUMMARY:
To review current Emergency Department procedural sedation practices in the community hospital setting and the associated drugs used (class of anesthetic and mode of administration). The ultimate goal of this investigation is to determine the need for a new analgesic/anesthesia drug and to compare the outcomes of a new drug within the same community Emergency Department setting. In particular, this may present a future opportunity to evaluate Penthrox (methoxyflurane) as a viable alternative for procedural sedation and analgesia in Canadian Emergency Departments.

DETAILED DESCRIPTION:
Procedural sedation is a common practice in the Emergency Department setting. The purpose of procedural sedation is to provide adequate pain relief to patients undergoing an emergent procedure. As a result, the time to the patient's symptom relief, the degree of side effects and the duration of action of the medication are all critical to selecting an appropriate sedative and/or analgesic.

The community hospital setting may present unique challenges to successfully administering procedural sedation techniques. Funding and resource allocation can limit patient access to timely sedation/analgesia. This can be compounded by prolonged stays in the Emergency Department for recovery and/or complications.

The current recommendations for 'Procedural Sedation and Analgesia in the Emergency Department' outlines recommended medications and policies for adults and children undergoing procedural sedation1,2. While a number of cohort and retrospective analyses have been done in a variety of research settings, the role for oral or intranasal anesthesia has not been adequately explored in ED settings. The initial phase of this research proposal will identify current local practices through chart review analysis collected over the last year. Subsequent research questions might include a comparative analysis of the current procedural sedation techniques compared to medications administered orally or by inhalation. This may have considerable future benefit to patient satisfaction and clinical outcomes, as well as resource and operational outcomes in the Emergency Department.

Hypothesis

To identify interventions requiring procedural sedation and the medication commonly used in a Canadian community emergency department (ED). Using standardized medical record review methods, primary clinical patient indicators, safety outcomes and secondary ED operational outcomes will be reviewed.3

Study Design

This retrospective chart review will be obtained from data of patients who have registered in the Welland County General Hospital (WHS) from the dates of January 2017 -December 2018. This timeframe should capture a sample size of ~300 patients.

Patients will be included in our study if they have received conscious sedation for a diagnostic or therapeutic procedure in the emergency department. They will be identified through review of billing records for anesthesia codes. Medical records, specifically physician procedural sedation records and nursing documentation, will be our main resources for data extraction. The investigators will describe and quantify the procedures requiring conscious sedation and identify the medication (and route) used, using a standardized data abstraction tool to be created from international ED PSA guidelines.1,2 Primary outcome measures will include ED PSA indications, pre-procedural assessments (medical comorbidities, difficult airway predictors, other safety factors), medications used, sedation failures/use of rescue medications, procedural successes or failures, post-PSA assessments, PSA recovery and patient disposition. Further stratification by age and other demographic features will help us better understand trends between the adult and pediatric population.

Patients requiring anaesthesia for the purpose of intubation and ventilator support will be excluded from this study.

Our secondary outcomes involve resource utilization and complications. Duration of procedure and time to discharge will be measured. Data on adverse outcomes and unplanned admission rates will also be collected. Adverse outcomes of interest will be vomiting, medication for blood pressure support, dysrhythmias, unanticipated intubation, laryngospasm, pulse oximetry less than 90%, apnea requiring bag-valve-mask ventilation and death.

ELIGIBILITY:
Inclusion Criteria:

* patients who have registered in the Welland County General Hospital Emergency Department (WHS) from the dates of January 2017-December 2018.
* Patients who require procedural sedation in the Emergency Department

Exclusion Criteria:

- N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have registered in the Welland County General Hospital Emergency Department (WHS) from the dates of January 2017 -December 2018 and require procedural sedation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-11-30 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Procedural Sedation | 2 years
  Total number of patients requiring conscious sedation
Medication Use | 2 years
  The number and type of medications used during procedure
Pre Procedural Assessment Findings | 2 years
  ASA score, 3-3-2 Abnormality, Pre-procedure Fast, Mallampatie Class, Neck Obesity, Facial Hair
Sedation Failures and Use of Rescue Medications | 2 years
  Number of occurrences where sedation is inadequate for treatment and number/type of rescue medication used to achieve adequate sedation
Time of Discharge | 2 years
  Time of patient discharge or transfer from Emergency Department

SECONDARY OUTCOMES:
Length of time spent in Emergency Department | 2 years
Duration of Procedure and Time to discharge | 2 years
Number of Adverse Outcomes | 2 years
Rate of Hospital Admission | 2 years
Time from Triage to initiation of procedural sedation | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Niagara Health, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No